CLINICAL TRIAL: NCT02686879
Title: The Effect of Peripheral Defocus on Axial Growth and Modulation of Refractive Error in Hyperopes
Brief Title: Effect of Peripheral Defocus on Axial Growth in Hyperopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aston University (Other)
Collaborators: College of Optometrists (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 150-2015-IB
Record Dates: First submitted 2016-02-12; First posted 2016-02-22 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Hyperopia; Amblyopia; Anisohyperopia
Keywords: hyperopes; axial length; peripheral defocus
MeSH Terms: conditions — Hyperopia; Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Natural progession (No Intervention): Following the natural progression of axial growth and refractive error.
- Anisohyperopes - intervention eye (Experimental): The more hyperopic eye will be fitted with a centre-near multifocal contact lens
  Interventions: Device: Multifocal contact lenses
- Hyperopes (Experimental): Both eyes will be fitted with centre-near multifocal contact lenses.
  Interventions: Device: Multifocal contact lenses
- Anisohyperopes - fellow eye (Experimental): The less hyperopic eye will be fitted with a single vision contact lens if required.
  Interventions: Device: Single vision contact lenses

INTERVENTIONS:
Device: Multifocal contact lenses
  Arms: Anisohyperopes - intervention eye; Hyperopes
Device: Single vision contact lenses
  Arms: Anisohyperopes - fellow eye

SUMMARY:
Hyperopia, also known as farsightedness, is a common type of refractive error where distant objects may be seen more clearly than objects that are near.

Hyperopia is a known risk factor for amblyopia, (lazy eye), which may occur as a result of a squint (turn), or due to different levels of hyperopia between each eye (anisohyperopia).

Hyperopia and anisohyperopia often persist into adulthood resulting in impairment to binocular vision. Current management involves prescribing spectacles or contact lenses to correct the hyperopia in each eye, usually as a lifelong intervention.

In recent years there has been a great deal of interest in delaying progression of myopia (short-sightedness) by slowing down the growth of the eye using a particular type of contact lens termed a centre-distance multifocal design. There have been some encouraging results in this area to date.

The proposed study here would explore the use of centre-near multifocal design contact lenses to encourage growth of the eye, thereby reducing hyperopia. There are three elements to the programme of research:

1. The natural progression of axial growth and refractive error will be measured in hyperopic and anisohyperopic subjects aged between 5 and 19. In other words, the natural growth of the eye will be followed without any intervention
2. As a paired eye control study anisohyperopes aged between 8 and 15 will be fitted with a centre-near multifocal design contact lens in their more hyperopic eye and a single vision contact lens in the fellow eye, if required. The progression of axial growth and refractive error will be measured and compared in each eye
3. Subjects' aged between 8 and 15 with similar levels of hyperopia in each eye will be fitted with centre-near multifocal design contact lenses in each eye. The progression of axial growth and refractive error will be measured and compared to subjects in the natural progression study

DETAILED DESCRIPTION:
Currently, hyperopia receives much less research attention than myopia even though the impact of moderate to high levels of hyperopia especially in one eye (anisohyperopia) can lead to amblyopia if not corrected fully at a young age. Hyperopia occurs as a consequence of insufficient ocular growth and a failure to emmetropise (reach the expected normal level) in childhood with the majority of hyperopic refractive errors resulting from an eye that is too short for its refractive power. In anisohyperopia it is unclear why one eye may remain hyperopic while the fellow eye grows towards an emmetropic state. Studies on animals have suggested that manipulating peripheral defocus through optical means while simultaneously providing correct axial focus can either discourage or encourage axial growth to effectively treat myopia or hyperopia respectively. Recent research has established that progression of myopia and axial growth can be significantly reduced in children and adolescents through the use of bifocal or multifocal contact lenses.

The optometrist has a central role in the clinical management of refractive error in children and in the application of future modalities that may modify the development of ametropia. The following proposal, therefore, presents a programme of work that is both relevant to the optometrist and novel in hyperopia research. By combining assessment of ocular biometry, monitoring of normal growth rates, an intervention study using bifocal contact lenses in children will be the first to provide new data on whether human eyes can be stimulated to grow in response to a specific type of defocus. Consequently the research will offer a new perspective on the management of hyperopia and anisohyperopia. The findings will offer a potential new approach towards amblyopia treatment in children and insight into a strategy for optimal correction to encourage axial growth in hyperopia.

There will be three elements to the proposed programme of research:

* Refractive error and axial growth will be followed over a three year period in hyperopic and anisohyperopic subjects aged between 5 and 19 years old to gain understanding of natural progression of these parameters in the specified cohort
* Simultaneous vision bifocal/mulitfocal soft contact lenses will be used to encourage axial growth in hyperopic children and adolescents with axial hyperopia in an effort to reduce hyperopia. The bifocal centre near design contact lenses will be prescribed to provide for clear central vision at both distance and near thus exposing the retina to peripheral hyperopic defocus from the distance zone
* This concept will also be applied to anisometropes as they represent a unique example of ocular development, where the two eyes of an individual, with an identical genetic background and seemingly subject to identical environmental influences, can grow asymmetrically to produce significantly different refractive errors. This correction and manipulation strategy has the potential to be applied to the more hyperopic eye to encourage eye growth and reduction of hyperopia with associated benefits of improved binocular vision and stereopsis.

For the natural progression study healthy hyperopic children and adolescents aged between 5 and 19 years of age will be recruited via the researcher's optometry practices and Aston University optometry clinic. The growth and visual characteristics of the eyes will be followed over time without any intervention by the research team. Following consent, at the initial visit, all participants will undergo a number of visual assessments including measurement of the axial length of the eye, focusing ability over a range of distances, eye muscle balance, vision at a range of different contrasts, pupil size and quality of stereovision and objective assessment of the crystalline lens parameters. Measures of the participant's spectacle prescription by objective and subjective means will also be undertaken following the instillation of eye drops to relax the muscles of the eye and to dilate the pupils. The eye drops will take around 40 minutes to work with the pupils returning to normal size after approximately 24 hours. The majority of these assessments are similar to those undertaken during a routine eye examination. The height of the subjects will also be taken at baseline and at six monthly intervals throughout the study. Parents and children will also be asked to complete a background questionnaire at this visit. The first visit is expected to last around 90 minutes. Participants will be reviewed every six months over a period of three years where the measures taken at baseline will be repeated. Instillation of eye drops to dilate the pupils and relax the eye muscles will be used on alternate visits.

For the intervention study, at the initial visit all participants will undergo a number of visual assessments including measurement of the shape and length of the eye, focusing ability over a range of distances, eye muscle balance, vision at a range of different contrasts, pupil size and quality of stereovision. Measures of the participant's spectacle prescription by objective and subjective means will also be undertaken following the instillation of eye drops to relax the muscles of the eye and to dilate the pupils. Subjects in the intervention groups will be reassessed after a period of six months to establish a measure of natural eye growth prior to being fitted with contact lenses. Parents and children will also be asked to complete a background questionnaire at this visit. The first visit is expected to last around 90 minutes.

The second visit for the intervention group will be to assess the individual's suitability for contact lens wear using a microscope. The participant and parent will be instructed on how to insert, remove and care for their contact lenses. The fitting of the contact lenses and level of vision will be assessed. For the anisohyperopes, the more hyperopic eye will be fitted with a commercially available soft multifocal contact lens and the less hyperopic eye will be fitted with a soft single vision contact lens. Subjects with similar levels of hyperopia in each eye will be fitted with commercially available soft multifocal contact lenses in both eyes. The participant will then be issued with a supply of contact lenses along with commercially produced instruction guides on caring for their contact lenses. The second visit is expected to last around 90 minutes.

The child may need to attend for unscheduled visits if any problems arise during the early stages of contact lens wear. Otherwise they will be reviewed at one to two weeks after the dispensing visit and also one month later for routine contact lens aftercare appointments.

Participants in the intervention groups will be reviewed at 6, 12, 18 and 24 months after the dispensing visit. During these visits the majority of measurements undertaken during the initial assessment will be repeated along with routine contact lens aftercare. Eye drops to relax the eye muscles and dilate the pupils will be instilled at the 12 and 24 month visits. For the anisohyperopic subjects, if the level of hyperopia in the more hyperopic eye reduces to a level that matches the less hyperopic eye then the intervention will be stopped. For the non-anisohyperopic subjects, the intervention will be stopped when the refractive error has reached a mean spherical error of +0.50D. At the end of an intervention period of 24 months the participants will be assessed after a period of 6 months to assess the growth of their eyes post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 5 and 19 years at the initial examination for the natural progression arm
* Aged between 8 and 15 years at the initial examination for the intervention arms
* Parents must have read, understood and signed informed consent form
* Participants must have read, understood and signed assent form
* Participants in the intervention groups agree to wear the prescribed contact lenses for a minimum of 10 hours per day, at least 6 days per week for the 2-year duration of the intervention period
* Be in good general health with no contraindications to contact lens wear
* Maximum manifest spherical refractive error of +6.00D
* Maximum manifest cylindrical refractive error of -1.00D
* Minimum anisometropia of 1.25D in the anisohyperopic group (mean spherical error)
* Maximum anisometropia of 1.00D in the non-anisohyperopic group (mean spherical error)
* Minimum mean spherical refractive error of +2.00D in the more hyperopic eye
* Be competent at handling contact lenses and understand the instructions given to ensure safe wear.

Exclusion Criteria• Previous contact lens wear

* Participating within another clinical study (even if it is only an observational study?)
* Regular use of medication to treat ocular conditions
* Current use of systemic medication that may impact upon successful contact lens wear or affect focusing ability
* Known ocular or systemic disease
* Findings identified during contact lens assessment that would preclude contact lens wear.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2022-02 (Actual)

PRIMARY OUTCOMES:
Measurement in axial length change in mm | Three years
  Axial length measured at baseline. Intervention introduced six months after baseline measures for a period of two years. Final measures taken six months after removal of intervention. Total time frame of three years.

SECONDARY OUTCOMES:
Measurement of refractive change in dioptres | Three years
  Refraction measured at baseline. Intervention introduced six months after baseline measures for a period of two years. Final measures taken six months after removal of intervention. Total time frame of three years.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Eyesite Eyecare Centres, Coventry, Walsgrave
  - Aston University, Birmingham, West Midlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beasley IG, Davies LN, Logan NS. Effect of Peripheral Defocus on Axial Eye Growth and Modulation of Refractive Error in Hyperopes: Protocol for a Nonrandomized Clinical Trial. JMIR Res Protoc. 2018 Sep 5;7(9):e173. doi: 10.2196/resprot.9320. PMID 30185407